CLINICAL TRIAL: NCT03931928
Title: Genotype and Phenotype Guided Supplementation of TAMoxifen Standard Therapy With ENDOXifen in Breast Cancer Patients (TAMENDOX)
Brief Title: Genotype and Phenotype Guided Supplementation of TAMoxifen Standard Therapy With ENDOXifen in Breast Cancer Patients
Acronym: TAMENDOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Responsible Party: Principal Investigator, Matthias Schwab, Prof. Dr. med., Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKP275 / GBG91; 2016-000418-31 (EudraCT Number)
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; DCIS
Keywords: tamoxifen; endoxifen; endocrine receptor positive breast cancer; adjuvant therapy
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Group 1) (No Intervention): All patients receive Placebo
- Group 2 (Experimental): Patients will receive (Z)-endoxifen dosed according to CYP2D6 "genotype"
  Interventions: Drug: (Z)-Endoxifen supplementation according to genotype
- Group 3 (Experimental): Patients will receive (Z)-endoxifen dosed according to (Z)-endoxifen steady state plasma concentrations (phenotype) at screening
  Interventions: Drug: (Z)-Endoxifen supplementation according to plasma levels

INTERVENTIONS:
Drug: (Z)-Endoxifen supplementation according to genotype — Group 2: CYP2D6 genotype predicted intermediate metabolizer receive 1.5 mg, poor metabolizer receive 3 mg (Z)-Endoxifen and extensive or ultrarapid metabolizer receive 0 mg endoxifen (Placebo)
  Arms: Group 2
Drug: (Z)-Endoxifen supplementation according to plasma levels — Group 3: Patients will receive (Z)-endoxifen according to (Z)-endoxifen steady state plasma concentrations (phenotype) at screening (i.e. ≤ 15 nM receive 3 mg, > 15 and ≤ 25 nM receive 1.5 mg (Z)-Endoxifen and > 25 nM receive 0 mg (Placebo)
  Arms: Group 3

SUMMARY:
In hormone-receptor positive breast cancer or DCIS (ductal carcinoma in situ) tamoxifen remains an important treatment option for patients before menopause and those patients after menopause who cannot be treated with aromatase-inhibitors. Nonetheless, a considerable amount of patients suffer a relapse of their cancer while on treatment with tamoxifen. Tamoxifen is a drug that is metabolized to a variety of compounds by the human liver, and the most important antihormonally active metabolite is called (Z)-Endoxifen. It is known that patients who have a reduced or absent activity of the drug-metabolizing enzyme CYP2D6 have lower levels of (Z)-Endoxifen. Furthermore, it has been observed that patients on tamoxifen therapy who have absent CYP2D6 activity are at a 2-fold increased risk for disease recurrence, and patients with lower CYP2D6 compared to patients with normal CYP2D6 activity still have a 1.4-fold increased risk for disease recurrence.

This trial will include patients who are already on tamoxifen therapy for at least 3 months and is designed to show that in patients with absent or low CYP2D6 activity, (Z)-Endoxifen supplementation - that is giving (Z)-Endoxifen in addition to tamoxifen for the study period of 42 days - can increase blood levels of (Z)-Endoxifen to therapeutic concentrations. It is planned to included 504 patients in this blinded, randomized trial, which will have a placebo group (receiving no (Z)-Endoxifen) and two intervention groups that will receive 0, 1.5 or 3 mg (Z)-Endoxifen depending on their CYP2D6 genetics or their (Z)-Endoxifen levels at the start of the study.

The trial is not designed to evaluate outcome measures (that is recurrence or survival rates) of (Z)-Endoxifen supplementation in tamoxifen treated patients, but will document the safety of the combined administration of tamoxifen and (Z)-Endoxifen.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to study entry. The patient must be accessible for scheduled visits and treatment.
2. Pre- and postmenopausal women with ductal carcinoma in situ (DCIS) or early stage breast cancer. This includes stage I, IIA, IIB, and IIIA breast cancers.
3. ER+/PR+, ER+/PR- or ER-/PR+ receptor status. Criteria for endocrine sensitivity is ≥1% ER-positive or PR-positive tumor cells on immune-histochemical staining
4. Patients on standard tamoxifen monotherapy (20 mg/d) for at least three months or patients who had switched from AI to tamoxifen who are on tamoxifen treatment for at least three months
5. Age ≥ 18 years
6. Body mass index of 18.5 to 35.0 kg/m2
7. The Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
8. Absolute neutrophil count greater than or equal to 1 500/µL
9. Platelets greater than or equal to 100 000/µL
10. Total bilirubin within less than or equal to 1.5 times institutional upper limit of normal
11. AST/ALT less than or equal to 2.5 times institutional upper limit of normal
12. The subjects need to be either

    1. of non-childbearing potential (documented postmenopausal status, defined as no menses for 12 months without an alternative medical cause, or post hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or
    2. of childbearing potential (WOCBP) with negative serum pregnancy test (due to the known reproduction toxicity of tamoxifen found in preclinical studies, WOCBP need to use a highly effective non-hormonal contraception. These are copper IUDs, bilateral tubal ligation, a vasectomized partner (vasectomy at least three months prior to screening) or sexual abstinence. Male or female condoms with/ without spermicide or caps, diaphragms or sponges with spermicide are associated with a failure rate > 1% per year and are thus not sufficient during the intervention period.
13. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE version 5.0 Grade ≤ 2 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion)
14. Surgery and radiation therapy of the breast has to be completed upon study entry

Exclusion Criteria:

1. Subjects who are unable to understand written and verbal instructions
2. Locally advanced (Stadium IIIB or IIIC) or metastatic (Stage IV) breast cancer at the time of surgery
3. Ongoing chemotherapy and/or treatment with trastuzumab within the last three months; participation in another trial with any investigational/not-marketed drug within 3 months prior to baseline visit
4. Other active second malignancy
5. Invalid result of genotyping
6. Pregnancy
7. Breast feeding/lactation
8. Oral contraceptives containing estrogens and/or progesterones
9. Pathologic vaginal bleeding in pre-menopausal women or vaginal bleeding in post-menopausal patients
10. Current severe acute somatic or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in judgement of the investigator, would make the patient inappropriate for entry into this study.
11. Severe chronic cardiac or pulmonary disease (heart failure NYHA class 3 and 4), COPD GOLD C or D
12. Chronic or acute renal disease with a glomerular filtration rate < 60 ml/min/1.73 m2, and any patient on peritoneal dialysis or hemodialysis
13. Medical history of thromboembolism (deep vein thrombosis or pulmonary embolism)
14. QTc interval >0.47 sec at screening ECG
15. Concurrent treatment with strong to moderate inhibitors of CYP2D6 which may alter tamoxifen metabolism (Consortium on Breast Cancer Pharmacogenomics 2008):

    paroxetine, fluoxetine, bupropion, quinidine and duloxetine, diphenhydramine, thioridazine, amiodarone, cimetidine, sertraline
16. Known allergies against an ingredient of the investigational product or tamoxifen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with ductal carcinoma in situ (DCIS) or early stage breast cancer.
Enrollment: 356 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
(Z-)endoxifen plasma concentration > 32 nM | 42 days (-2 days/+7 days)
  The primary endpoint is reached if in one or both intervention groups, the proportion of patients with steady state (Z)-endoxifen plasma concentration > 32 nM is greater or equal to the proportion of patients in the control group that reaches steady state (Z)-endoxifen plasma concentration of > 32 nM

SECONDARY OUTCOMES:
Increase in steady state (Z)-endoxifen concentration | 42 days (-2 days/+7 days)
  Increase in steady state (Z)-endoxifen concentration from baseline to end of intervention (Visit 3) in patients with or without supplementation of (Z)-endoxifen
Change in steady state plasma concentrations of tamoxifen, desmethyltamoxifen, 4-hydroxytamoxifen and other tamoxifen metabolites following (Z-)endoxifen supplementation | 42 days (-2 days/+7 days)
  Assessment of steady state plasma concentrations of tamoxifen, desmethyltamoxifen, 4-hydroxytamoxifen, and other tamoxifen metabolites following (Z)-endoxifen supplementation for 6 weeks

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | AE/SAE occurring while the subject is on IMP, or within 30 days of the patient's last dose of IMP
  All AE/SAE occuring in the intervention period will descriptively reported

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Schwab, Prof. Dr., Principal Investigator — Margarete Fischer-Bosch-Institute of Clinical Pharmacology
Locations (40):
- Germany (40):
  - Gemeinschaftspraxis für Gynäkologie und Geburtshilfe Salzgitter, Salzgitter, Albert-Schweitzer-Straße 18
  - Zentralklinikum Suhl, Klinik für Frauenheilkunde/Geburtsmedizin, Zentrum für klinische Studien, Suhl, Albert-Schweitzer-Straße 2
  - Rems-Murr-Klinikum-Winnenden, Frauenklinik, Winnenden, Am Jakobsweg 1
  - Robert-Bosch-Krankenhaus, Stuttgart, Auerbachstr. 112
  - Onkologische Gemeinschaftspraxis Hildesheim, Gynäkologie, Hildesheim, Bahnhofsplatz 5
  - Johanniter-Krankenhaus Stendal, Klinik für Frauenheilkunde und Geburtshilfe, Stendal, Bahnhofstr. 24-26
  - Klinikum Magdeburg, Klinik für Hämatologie/Onkologie, Magdeburg, Birkenallee 34
  - Klinikum Memmingen, Brustzentrum, Memmingen, Bismarckstraße 23
  - Klinikum am Bruderwald Bamberg, Hämatologie/Internistische Onkologie, Bamberg, Buger Straße 80
  - MVZ am Klinikum am Bruderwald Bamberg, Bamberg, Buger Straße 80
  - Universitätsfrauenklinik Tübingen, Tübingen, Calwer Straße 7
  - Helios Klinikum Gifhorn, Interdisziplinäres Brustzentrum, Gifhorn, Campus 6
  - ViDiA Christliche Kliniken Karlsruhe, Frauenklinik, Karlsruhe, Diakonissenstr.28
  - Klinikum Quedlinburg, Frauenklinik, Quedlinburg, Ditfurter Weg 24
  - Klinikum Höchst Frankfurt am Main, Klinik für Gynäkologie und Geburtshilfe, Frankfurt am Main, Gotenstr. 6-8
  - Evangelisches Diakonie-Krankenhaus Bremen, Frauenklinik, Bremen, Gröpelinger Heerstraße 406-408
  - Onkologische Gemeinschaftspraxis Brudler-Heinrich-Bangerter Augsburg, Augsburg, Halderstraße 29
  - medius Klinik Ostfildern-Ruit, Brustzentrum, Ostfildern, Hedelfingerstraße 166
  - Helios Universitätsklinikum Wuppertal GmbH, Brustzentrum, Wuppertal, Heusnerstraße 40
  - Klinikum Esslingen, Klinik für Frauenheilkunde, Brustzentrum, Esslingen am Neckar, Hirschlandstraße 97
  - SRH Kliniken Sigmaringen, Gynäkologie und Geburtshilfe, Sigmaringen, Hohenzollerstr. 40
  - Harz-Klinikum Wernigerode, Abteilung Gynäkologie und Geburtshilfe, Wernigerode, Ilsenburger Straße 15
  - Klinikum Passau, Gynäkologische Onkologie, Passau, Innstraße 76
  - St. Johannes Hospital Dortmund, Klinische Forschung, Dortmund, Johannesstraße 9-17
  - Marienhospital Bottrop, Klinik für Gynäkologie und Geburtshilfe, Bottrop, Josef-Albers-Straße 70
  - Universitätsfrauenklinik Mainz, Klinik und Poliklinik für Geburtshilfe und Frauenheilkunde, Mainz, Langenbeckstr. 1
  - Onkozentrum Dresden, Fachärzte für Innere Medizin, Hämatologie und Internistische Onkologie, Dresden, Leipziger Straße 120
  - HELIOS Dr. Horst Schmidt Kliniken Wiesbaden, Klinik für Gynäkologie und gyn. Onkologie, Wiesbaden, Ludwig-Erhard-Straße 100
  - Luisenkrankenhaus Düsseldorf GmbH & Co. KG, Brustzentrum, Düsseldorf, Luise-Rainer-Straße 6-10
  - Marienhospital Witten, Brustzentrum, Witten, Marienplatz 2
  - Städtisches Klinikum Karlsruhe, Frauenklinik, Karlsruhe, Moltkestr. 90
  - Kliniken der Stadt Köln, Brustzentrum Köln-Holweide, Cologne, Neufelder Straße 32
  - Diakonissen-Krankenhaus Speyer, Klinik für Gynäkologie und Geburtshilfe, Speyer, Paul-Egell-Straße 33
  - Klinikum Ludwigsburg, Frauenklinik, Ludwigsburg, Posilipostraße 4
  - DRK Kliniken Berlin-Köpenick, Frauenklinik, Köpenick, Salvador-Allende-Straße 2-8
  - MVZ Eggenfelden, Gynäkologische Onkologie, Eggenfelden, Schellenbruckerstr. 15
  - Klinikum am Steinenberg Reutlingen, Frauenklinik, Reutlingen, Steinenbergstr. 31
  - SRH Wald-Klinikum Gera GmbH, Klinik für Frauenheilkunde/Geburtsmedizin, Gera, Straße Des Friedens 122
  - Elisabeth Krankenhaus Kassel gGmbH, Brustzentrum, Kassel, Weinbergstr. 7
  - MVZ am Schlosssee Gifhorn, Gifhorn, Zur Allerwelle 4